CLINICAL TRIAL: NCT03255174
Title: A Prospective Study Evaluating the Safety and Effectiveness of EVARREST® Fibrin Sealant Patch in Controlling Mild or Moderate Hepatic Parenchyma or Soft Tissue Bleeding During Open Abdominal, Retroperitoneal, Pelvic and Thoracic (Non-cardiac) Surgery in Pediatric Patients
Brief Title: The EVARREST® Pediatric Mild or Moderate Liver and Soft Tissue Bleeding Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIOS-16-001
Record Dates: First submitted 2017-07-13; First posted 2017-08-21 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Controlling Mild to Moderate Bleeding During Surgery
Keywords: Bleeding, hemostasis, re-bleeding, hemostatic
MeSH Terms: conditions — Hemorrhage | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EVARREST® Fibrin Sealant Patch (Experimental): EVARREST Fibrin Sealant Patch is a sterile, bio-absorbable combination product consisting of two constituent parts- a flexible matrix and a coating of biological components (human plasma-derived fibrinogen and thrombin) embedded in a flexible composite patch component.
  Interventions: Biological: EVARREST® Fibrin Sealant Patch

INTERVENTIONS:
Biological: EVARREST® Fibrin Sealant Patch — EVARREST Fibrin Sealant Patch is a sterile, bio-absorbable combination product consisting of two constituent parts- a flexible matrix and a coating of biological components (human plasma-derived fibrinogen and thrombin) embedded in a flexible composite patch component.
  Other Names: EVARREST

SUMMARY:
The objective of this study is to evaluate the safety and hemostatic effectiveness of EVARREST as an adjunct to controlling mild to moderate soft hepatic parenchyma or soft tissue bleeding during open hepatic, abdominal, pelvic, retroperitoneal, and thoracic (non-cardiac) surgery in pediatric population.

DETAILED DESCRIPTION:
This is an open-label, multicenter, single-arm study evaluating the safety and effectiveness of EVARREST in controlling mild or moderate bleeding in hepatic parenchyma or soft tissue for which standard methods of achieving hemostasis are ineffective or impractical.

Eligible subjects will be treated with EVARREST. Subjects will be followed post-operatively through discharge and at 30 days (+/-14 days) post-surgery.

At least thirty-five pediatric subjects with an appropriate mild or moderate bleeding target bleeding site (TBS) will be enrolled in this study. The age of the subjects enrolled in the study will be from 1 month to less than (<) 18 years. This will include a minimum of 4 subjects aged 1 month (greater than or equal to [>=] 28 days from birth) to <1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric subjects aged ≥28 days (≥1 month) to <18 years, requiring non-emergent open hepatic, abdominal, retroperitoneal, pelvic or thoracic (non-cardiac) surgical procedures; i) A minimum of 4 subjects to be enrolled will be aged ≥28 days to <1 year
2. The subject's parent/legal guardian must be willing to give permission for the subject to participate in the trial, and provide written Informed Consent for the subject. In addition, assent must be obtained from pediatric subjects who possess the intellectual and emotional ability to comprehend the concepts involved in the trial. If the pediatric subject is not able to provide assent (due to age, maturity and/or inability to intellectually and/or emotionally comprehend the trial), the parent/legal guardian's written Informed Consent for the subject will be acceptable for the subject to be included in the study.
3. Presence of an appropriate mild or moderate bleeding soft tissue or hepatic parenchyma Target Bleeding Site (TBS) identified intra-operatively by the surgeon;
4. Ability to firmly press trial treatment at TBS until 4 minutes after TBS identification.

Exclusion Criteria:

1. Subjects with known intolerance to blood products or to one of the components of the study product or is unwilling to receive blood products;
2. Female subjects, of childbearing age (i.e. adolescent), who are pregnant or nursing;
3. Subject is currently participating or plan to participate in any other investigational device or drug study without prior approval from the Sponsor;
4. Subjects who are known, current alcohol and/or drug abusers
5. Subjects admitted for trauma surgery
6. Subjects with any pre or intra-operative findings identified by the surgeon that may preclude conduct of the study procedure
7. Subjects that have received a COVID-19 vaccine either 4 weeks prior to surgery or scheduled to receive COVID-19 vaccine within the 30-day follow-up period
8. Subject with TBS in an actively infected field (Class III Contaminated or Class IV Dirty or Infected)
9. TBS is from large defects in arteries or veins where the injured vascular wall requires repair with maintenance of vessel patency and which would result in persistent exposure of EVARREST to blood flow and pressure during healing and absorption of the product
10. TBS with major arterial bleeding requiring suture or mechanical ligation;
11. Bleeding site is in, around, or in proximity to foramina in bone, or areas of bony confine.

Ages: 28 Days to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Absolute time to hemostasis | Intraoperative from TBS identification to the last moment in time at which no detectable bleeding at the TBS is observed
  The absolute time to hemostasis, defined as the absolute time elapsed from TBS identification to the last moment in time at which detectable bleeding at the TBS is observed.

SECONDARY OUTCOMES:
Hemostatic success at 4 minutes | Intraoperative, 4 minutes after TBS identification
  Proportion of subjects achieving hemostatic success at 4 minutes following Target Bleeding Site (TBS) identification and no bleeding requiring treatment at the TBS any time prior to final fascial closure.
Hemostatic success at 10 minutes | Intraoperative, 10 minutes after TBS identification
  Proportion of subjects achieving hemostatic success at 10 minutes following TBS identification and no bleeding requiring treatment at the TBS any time prior to final fascial closure.
No re-bleeding at the TBS | Intraoperative, from TBS identification to final fascial closure
  Proportion of subjects with no re-bleeding at the TBS.
Incidence of adverse events that are potentially related to bleeding at the TBS | Intraoperative to 30 (+/- 14) days
  Incidence of adverse events that are potentially related to bleeding at the TBS.
Incidence of adverse events that are potentially related to thrombotic events | Intraoperative to 30 (+/- 14) days
  Incidence of adverse events that are potentially related to thrombotic events.
Incidence of re-treatment at the TBS | Intraoperative, from TBS identification to final fascial closure
Incidence of Adverse Events | Intraoperative to 30 (+/- 14) days
Number of Participants with Abnormalities in Clinical Laboratory Tests | Intraoperative to 30 days
  Number of participants with abnormalities in clinical laboratory tests (hemoglobin, hematocrit, and platelets) will be reported.
Number of Participants with Estimated Intraoperative Blood Loss | Intraoperative to 30 days
  Number of participants with estimated intraoperative blood loss will be reported.
Number of Participants with Blood products Transfused | Intraoperative to 30 days
  Number of participants with blood products transfused will be reported.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - University of Alabama Hospital, Birmingham, Alabama
  - icahn School of Medicine at Mt Sinai, New York, New York
- United Kingdom (3):
  - Birmingham Chrildren's Hospital, Birmingham
  - Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Southampton University Hospital, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Efficacy and safety results related to the primary and secondary endpoints